CLINICAL TRIAL: NCT03185884
Title: An Evaluation of Carbohydrates and Children
Brief Title: Carbohydrates and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: AL25
Record Dates: First submitted 2017-05-22; First posted 2017-06-14 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Carbohydrate Metabolism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): - 237 ml beverage; consumed once per test visit
  Interventions: Other: Control
- Experimental (Experimental): - 237 ml beverage; consumed once per test visit
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Control — control carbohydrate blend
  Arms: Control
Other: Experimental — experimental carbohydrate blend
  Arms: Experimental

SUMMARY:
This study will evaluate the impact of test carbohydrate blends on fat and carbohydrate oxidation, glucose, insulin and hunger scores in pre-adolescent boys and girls.

ELIGIBILITY:
Inclusion Criteria:

* Male 9 -13 years of age, or female 9- 10 years of age
* Tanner stage 1
* Subject was born full term
* Subject was born normal weight
* Subject passes the Physical Activity Readiness Questionnaire
* Body mass index >5th percentile and <95th percentile for age and gender
* Subject has voluntarily signed and dated a youth assent document

Exclusion Criteria:

* History of metabolic. endocrine, or hyperactivity disorders
* Allergy or intolerance to any ingredient found in the study products
* Participation in a concomitant trial of a non-registered drug or that otherwise conflicts with this study

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2017-08-12 (Actual); Study Completion 2017-08-12 (Actual)

PRIMARY OUTCOMES:
Energy Utilization | Study Visits 1 to 2 (1- 14 days)
  Calculated by Indirect Calorimetry using volume of oxygen consumed (liters/minute) and the volume of carbon dioxide expired (liters/minute).

SECONDARY OUTCOMES:
Hunger Assessment | Study Visits 1 to 2 (1- 14 days)
  Visual analog scale (units on a scale)
Blood Measurements - Glucose | Study Visits 1 to 2 (1- 14 days)
  mg/dl
Blood Measurements - Insulin | Study Visits 1 to 2 (1- 14 days)
  IU

CONTACTS AND LOCATIONS:
Overall Officials: Vikkie Mustad, PhD, Study Chair — Abbott Nutrition
Locations (1):
- University of Nebraska-Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gillen ZM, Mustad VA, Shoemaker ME, Mckay BD, Leutzinger TJ, Lopez-Pedrosa JM, Rueda R, Cramer JT. Impact of slow versus rapid digesting carbohydrates on substrate oxidation in pre-pubertal children: A randomized crossover trial. Clin Nutr. 2021 Jun;40(6):3718-3728. doi: 10.1016/j.clnu.2021.05.004. Epub 2021 May 11. PMID 34130017
- [Derived] Shoemaker ME, Gillen ZM, Mckay BD, Leutzinger TJ, Mustad VA, Cramer JT. Endogenous versus exogenous carbohydrate oxidation measured by stable isotopes in pre-pubescent children plus 13C abundances in foods consumed three days prior. Metabol Open. 2020 Jul 15;7:100041. doi: 10.1016/j.metop.2020.100041. eCollection 2020 Sep. PMID 32812942